CLINICAL TRIAL: NCT03278171
Title: Early Detection of Patients at Risk of Developing a Post-traumatic Stress Disorder After a Stay in Intensive Care Unit
Acronym: STRESSREA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0462
Record Dates: First submitted 2017-09-05; First posted 2017-09-11 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2017-09

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in intensive care unit: Cohort of patients leaving intensive care unit after a stay of more than 72 hours
  Interventions: Behavioral: Impact Event Scale Revisited

INTERVENTIONS:
Behavioral: Impact Event Scale Revisited — Evaluating the ability of the Impact Event Scale -Revisited within 8 days following the intensive care unit exit to predict a post-traumatic stress disorder at 3 months (Impact Event Scale -Revisited score strictly greater than 34)

SUMMARY:
Post-traumatic stress disorder (PTSD) is a psychiatric pathology noticed in the DSM-5, in troubles due to a traumatism or a stress factor and appearing at least 1 month after confrontation with trauma. This trouble can become chronic, and be the source of psychiatric and somatic comorbidities, which themselves have personal, professional and economic consequences at the level of the individual and society.

Some studies looked at the psychological effects induced by a stay in intensive care unit (ICU) since few years. The emergence of PTSD in these patients has been described, with an incidence varying from 4% to 60%.

The literature is contradictory about identified risk factors for PTSD. It's not possible to design a screening of these patients actually, only focused on the risk factors. It has been shown that the presence of acute stress trouble (presence of symptoms during the first month after the traumatism) was a risk factor for PTSD. Early detection of acute stress disorder could be a way to screen risk of emergence of a post-intensive care PTSD. Post-intensive care consultations have been done at 6 months, but not systematically. Only few symptoms are looked for and a sizable part of this population were not being followed probably due to a non-diagnosed-PTSD. In case of the emergence of a post-intensive care PTSD, those patients will never be diagnosed and treated, favoring all complications linked to this trouble.

Associated with other factors, IES-R (Impact Event Scale Revisited) at the ICU exit would permit an exhaustive screening of patients at risk for PTSD and could permit to propose them an adapted care and then limit the emergence of PTSD and its consequences..

In this study, the investigators will screen acute stress symptoms within 8 days following the ICU's exit, using the IES-R, in order to evaluate his ability to predict the emergence of a PTSD at three months. IES-R is an auto-questionnaire, easy and fast with good psychometrics capacities for PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old leaving an intensive care unit after a stay of more than 72 hours, in one of the medical and surgical intensive care units of the E Herriot Hospital
* Patient having given his agreement to participate in this study

Exclusion Criteria:

* Patient not understanding French language
* Confused patient (clinical assessment)
* Patient under protection measure or deprived from his rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People over 18 years old, staying more than 72 hours in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Impact Event Scale Revisited | 3 months
  Impact Event Scale Revisited (IES-R) will be carried out by a psychiatry clinician within 8 days following the intensive care unit in order to evaluate his ability to predict the emergence of a PTSD at three months. IES-R is an auto-questionnaire, easy and fast with good psychometrics capacities for PTSD.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatrie des urgences, Hôpital Edouard Herriot, Lyon, France

IPD SHARING:
Plan to Share IPD: No